CLINICAL TRIAL: NCT06624579
Title: Prognostic Value of Confocal Endomicroscopy in Ulcerative Colitis: the CONF-UC Study
Acronym: CONF-UC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FEDERICA FURFARO (Other)
Responsible Party: Sponsor-Investigator, FEDERICA FURFARO, PhD, MD, IRCCS Ospedale San Raffaele
Organization: IRCCS Ospedale San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRCCS SAN RAFAEL HOSPITAL
Record Dates: First submitted 2024-08-21; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: 26 adult subjects with moderate-to-severe active (defined as having patient-reported outcomes, PRO > 2), left-sided or extensive UC, requiring small molecules therapy according to the standards of care (ECCO guidelines) and performing routine investigations with Colonoscopy before starting appropriate therapy, according to the current standard of care indications and ECCO guidelines.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- confocal endomicroscopy (Other): Endoscopic confocal microscopy with fluorescein injection is a medical imaging technique that combines endoscopy with confocal microscopy and the injection of fluorescein, a fluorescent dye.
  During colonoscopy or rettosigmoidoscopy, confocal microscopy is used, which provides high-resolution images of tissues at a cellular level. This technology uses a thin probe with a laser light source and a detection system to analyze specific layers of tissue. During the examination, a solution of fluorescein is injected into the patient's peripheric vein. Fluorescein is a dye that binds to cellular structures, making them fluorescent when exposed to laser light. This allows to visualize cellular details in real-time during endoscopy
  Interventions: Procedure: confocal endomicroscopy

INTERVENTIONS:
Procedure: confocal endomicroscopy — The study incorporates confocal endomicroscopy as an additional diagnostic modality for assessing barrier dysfunction and treatment response in UC patients. Confocal endomicroscopy enables real-time visualization of mucosal changes at a cellular level during endoscopy, potentially enhancing the detection of treatment response and mucosal healing.

SUMMARY:
This study employs a prospective, single-center, interventional design to investigate the prognostic value of confocal endomicroscopy in assessing treatment response in ulcerative colitis (UC) patients receiving small molecules .

DETAILED DESCRIPTION:
The study incorporates confocal endomicroscopy as an additional diagnostic modality for assessing barrier dysfunction and treatment response in UC patients. Confocal endomicroscopy enables real-time visualization of mucosal changes at a cellular level during endoscopy, potentially enhancing the detection of treatment response and mucosal healing.

Eligible patients will undergo baseline assessment, including clinical evaluation, partial Mayo score calculation, endoscopic evaluation, biopsies with histological evaluation and confocal endomicroscopy. Follow-up assessments will be conducted at 8 weeks and 6 months after initiating therapy with small molecules .

The study aims to enroll a sample size of 26 UC patients to pilot the feasibility and utility of confocal endomicroscopy in assessing barrier dysfunction and treatment response.

ELIGIBILITY:
Inclusion Criteria:

1. Established diagnosis of UC since at least 12 weeks prior to inclusion
2. Age ≥ 18 years
3. Any gender/sex
4. Active disease consistent with indication to start with Small molecules (defined as Mayo endoscopic score (MES) ≥ 1, partial Mayo score ≥ 3 (with at least rectal bleeding score of 1 and bowel movements score of 1)
5. No contraindications to endoscopy or confocal exam
6. Ability to understand and to comply with the study procedure and sign an informed consent form

Exclusion Criteria:

1. Subjects with an endoscopic Mayo sub-score at baseline <2;
2. Pregnancy
3. Subjects with any contraindication to any study procedure (included fluorescein allergy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Prognostic Value of Confocal Endomicroscopy in Ulcerative Colitis | at 8 weeks and 6 months to treatment initiation
  The study incorporates confocal endomicroscopy as an additional diagnostic modality for assessing barrier dysfunction and treatment response in UC patients. Confocal endomicroscopy enables real-time visualization of mucosal changes at a cellular level during endoscopy, potentially enhancing the detection of treatment response and mucosal healing.